CLINICAL TRIAL: NCT00337337
Title: Effect of Reconstitute Multiple Grain on Glucose and Lipid Metabolism in Patients With Type 2 Diabetes
Brief Title: Multiple Grain in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCKU-94-032
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; rice; fiber
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Behavioral: Multiple grain
Behavioral: Ordinary Asian- rice

SUMMARY:
We aim to investigate the beneficial effect of adding grain fiber to daily rice meal in type 2 diabetic patients. We anticipate this intervention will improve glycemia and lipid profile in these patients.

DETAILED DESCRIPTION:
Resistance of insulin-mediated glucose transport is a fundamental early defect in the pathogenesis of type 2 diabetes mellitus (DM). It has been found that high fiber concentration in meal is frequently associated with low GI. In many single-blind cross-over study, short term consumption of high fiber meal has been shown to enhance postprandial insulin sensitivity in healthy subjects. We presume that increasing daily consumption of fiber would improve the insulin resistance and therefor glycemic parameters patients with DM. Patients with type 2 diabetes with stable dose of hypoglycemic medication control will be recruited, two types of meals will be given, type A is a general Asian rice-meal and type B consists of the same rice with multiple-grain-fiber added. Both type of meals will be consumed for 3 months by each patients.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent adults of either sex with age 30-75 years old
* Patients have type 2 diabetes mellitus diagnosed after 25 years of age
* Patients have been in inadequate but stable glycemic control by diet. Inadequate glycemic control isdefined as: HbA1c 7.1-11.0%
* Patients have signed the written informed consent.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus
* Patients with alcohol, drugs or medications abuse considered by the investigator
* Patients with impaired liver function (AST, ALT>2.5× upper limit of normal)
* Patients with impaired kidney function (serum creatinine>3.0 mg/dl)
* Patients with emphysema or chronic bronchitis
* Patients with hepatic cirrhosis
* Patients with chronic intestinal diseases related to marked disorders of digestion or absorption
* Patients participated investigational drug trial within 1 month before entering this study
* Patients with any other serious diseases considered by the investigator not in the condition to enter the trial

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2007-02

PRIMARY OUTCOMES:
Changes in glycemic parameters including fasting plasma glucose, postprandial plasma glucose, insulin sensitivity and lipid profile

SECONDARY OUTCOMES:
Changes in body weight
Acceptabiliy and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: T-J Wu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan